CLINICAL TRIAL: NCT02630446
Title: Effectiveness and Cost-effectiveness of an In-home Respite Care Program to Support Informal Caregivers of People With Dementia: a Comparative Study
Brief Title: An In-home Respite Care Program to Support Informal Caregivers of People With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: InBev-Baillet Latour Fund (Unknown); Baluchon Alzheimer Belgium vzw (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E/01447/15
Record Dates: First submitted 2015-11-24; First posted 2015-12-15 (Estimated); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Dementia
Keywords: respite care; effectiveness; cost-effectiveness; support; caregiver; dementia; community-based
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- in-home respite care program (Experimental): During the respite care period, lasting at least five days, a trained or experienced care worker for persons with dementia takes over all caregiving tasks while the informal caregiver is absent. The care worker thus temporary moves into the house of the person with dementia. The care worker also writes down his/her observations in a diary as well as daily experiences and strategies on how to manage the difficult behaviors the caregivers listed before. So additionally to the provision of respite, this program also includes caregiver support and psycho-education. This support enables the caregiver to validate theirs perceptions, to learn how to deal with difficult behaviors and to feel understood by somebody.
  Interventions: Other: in-home respite care program
- standard dementia care (No Intervention): Control group receiving all types of standard dementia care except in-home respite care of the Baluchon type.

INTERVENTIONS:
Other: in-home respite care program — During the respite care period, lasting at least five days, a trained or experienced care worker for persons with dementia takes over all caregiving tasks while the informal caregiver is absent. The care worker thus temporary moves into the house of the person with dementia. The care worker also writes down his/her observations in a diary as well as daily experiences and strategies on how to manage the difficult behaviors the caregivers listed before. So additionally to the provision of respite, this program also includes caregiver support and psycho-education. This support enables the caregiver to validate theirs perceptions, to learn how to deal with difficult behaviors and to feel understood by somebody.
  Other Names: intervention group
  Arms: in-home respite care program

SUMMARY:
The general objective of this quasi-experimental study is to assess the effectiveness of an in-home respite care program compared to a control group not receiving the same type of in-home respite on the well-being of the caregiver, the care-recipient and on the healthcare system. The latter in terms of resource use, intention to institutionalize the care-recipient and time to nursing home placement.

A quasi-experimental study will be designed. The intervention group will consist of caregiver/care-recipient dyads receiving an in-home respite program called "Baluchonnage" and will be compared to a control group that doesn't receive "Baluchonnage". Comparison between the groups will be done by collecting health related and economic data. The trial will evaluate outcomes as well in the caregiver as in the care recipient (measured via the caregiver). The primary research outcome is caregiver burden. Secondary outcomes for caregivers are: health related quality of life and reactions to behavioral problems of the care-recipient. A secondary outcome related to the care-recipient is: frequency of behavioral problems. Secondary outcomes for the healthcare system are: intention to institutionalize the recipient into a nursing home and resource use of the recipient. Finally, in a follow up phase of the trial possible differences in time to nursing home placement will be measured (as well as burden and intention to institutionalize. Additionally, willingness to pay for "Baluchonnage" per day will be asked to the informal caregivers. Eventually, if the intervention is effective, modeled and trial based cost-effectiveness analyses will be undertaken in a separate economic evaluation plan.

DETAILED DESCRIPTION:
The in-home respite intervention group will receive in-home respite care also called "Baluchonnage". During that period, lasting at least five days (24/24hours), an internally trained or experienced care worker for persons with dementia takes over all caregiving tasks while the caregiver takes a break. This care worker also writes down his/her observations in a diary. The content of this diary enables the caregiver to validate their perceptions, provides strategies to deal with difficult situations, and let them feel that somebody can truly understand their daily challenges. The control group receives usual care (standard dementia care).

Participants of the in-home respite intervention group will be recruited by Baluchon staff when asking for a first or a new period of in-home respite care. First, Baluchon staff will describe the study to the dyads and ask them about their preparedness to participate. When they give their verbal consent contact information will be forwarded to the research team who will then contact them by phone. During this call a home visit will be planned to sign the informed consent and complete the baseline assessment. Participants in the control group will be recruited from several general practitioners spread over the different regions in Belgium. Potentially, in a later phase, control group participants will also be recruited via Memory Clinics in Belgium.

Similar to the recruitment of the intervention group, the physician will give some information about the study. When verbal consent to participate is given to the physician, caregivers will be contacted by phone by the research team to check eligibility. This will be done by listing different support strategies (including "Baluchonnage") and ask the caregiver if they would be interested to receive this type of support. Also previous use of Baluchonnage will be questioned because this is not allowed in the control group. When caregivers appear to be eligible the research team will plan a home visit to sign the informed consent and complete the baseline assessment.

Data collection of caregiver and care-recipient characteristics and research outcomes will be gathered at several assessment moments. The baseline assessment will be conducted during a home visit by a member of the research team. Background characteristics and baseline values of the research outcomes will be gathered during this assessment. For the intervention group this will be in the week preceding the respite period. For the control group this will take place after inclusion. A second assessment will be done in the intervention group two weeks after having the intervention. A third assessment moment will be done 6 months after inclusion and a last follow up assessment will be conducted after 12 months. To fulfill the assessments after the baseline assessment, caregivers will be contacted by telephone. All questionnaires will be available in Dutch and French for use in Belgium. When no valid translation of a certain questionnaire exists in Dutch or French for Belgium a back-forward translation method will be performed.

For caregivers the researchers will obtain the following background characteristics: age, gender, region, marital status, ethnicity, educational level, relationship with the care-recipient, employment status, living situation and time spent in caregiving. In both study groups the reason for (potential) use of respite will be asked. Earlier use of Baluchonnage will also be questioned to intervention group participants. Time spent in caregiving (measured twice) will be calculated using the RUD instrument (Resource Utilization in Dementia). For the care-recipient the following background characteristics will be collected at baseline: age, gender, marital status, ethnicity, region, National Registration Number, educational level, being on a waiting list for long-term nursing home placement, dementia-specific medication use, and severity of dementia. The National Registration Number of the person with dementia will be gathered. This will allow us to trace study participants in the IMA database (Intermutualistisch Agentschap) and gather information on resource use and date of placement in a nursing home over a longer time period than the trial. ADL (Activities of Daily Living) functioning will be measured using the Belgian Katz scale and severity of dementia with the Global Deterioration Scale. Both will be measured twice (baseline and after 6 months).

Sample size calculation is performed using SPSS SamplePower 3®. First, literature was searched to determine the needed effect size and standard deviation (SD) allowing to distinguish a statistical significant and clinical relevant difference in the primary outcome, i.e. burden. Based on the findings of a similar high quality intervention study an effect size of 0.4 was used in the analysis, which implies a difference of six points on the ZBI scale (Zarit Burden Interview), and a SD of 15. Also, an average drop-out rate of 20% was taken into account, a power of 80% and a significance level at 0.05. Based on these values a total of 124 caregiver/care-recipient dyads will be needed for the intervention group. To reduce selection-bias inherent to quasi-experimental studies an allocation ratio of 1:2 will be used to allow matching techniques. As a result 248 caregiver/care-recipient dyads will be needed in the control group.

When appropriate, i.e. if the intervention demonstrates an effect in the study endpoints, within-trial and modeled cost-effectiveness analyses will be conducted in a separate economic evaluation plan. First the analysis will be performed from the perspective of the health care payer taking into account direct health care costs for the government's health care budget (RIZIV/INAMI) as well as patients' co-payment. Assuming that policy makers would consider reimbursement of in-home respite in the future the daily cost of Baluchonnage will thus be included in the analyses. Alongside the costs of Baluchonnage other costs of healthcare resource use including hospital and community care will be included. Additionally, also a full societal viewpoint will be undertaken not only including potential health care costs for the health care budget and patients, but also all other direct and indirect costs for caregivers and patients. Because in this viewpoint everyone affected by the intervention should be considered, caregiver time and costs (i.e. time spent in caregiving and productivity loss) as well as resource use and costs of other sectors (f.e. food delivery) should be included. Based on the KCE (Belgian Health Care Knowledge Center) guidelines for health economic evaluations in Belgium future costs will be discounted at 3% and future QALY's at 1.5%. Health utilities or QALY's of caregivers from both intervention arms will be derived from the Belgian public preference list based on scores on the EQ-5D (general utility instrument). Decision analytic modeling will be carried out to extrapolate effects of the intervention found in the trial to a longer time horizon. The model will be based on results from the trial as well as existing data from literature. Assumptions, hypotheses and sources of information will be represented in a transparent and clear way. Finally, the model will be validated by experts.

Data on resources used by the care-recipient of each study group will be obtained by an adapted version of the RUD instrument at baseline and after six months inclusion. This RUD instrument attempts to include all resource use including: health care resource use containing hospital resources (in-patient and out-patient attendances,…) and community care resources (general practitioner visits, nurse visits,…), caregiver and patient resources (time spent in caregiver,…), and resource use in other sectors (social worker visits, home help visits,…). Duration and frequency of the used services will be multiplied by each unit cost of the corresponding service. These unit costs will be obtained from the Belgian Reimbursement scheme using standard fees for regularly insured patients and other publicly available sources. Time spent in caregiving will be calculated at baseline and after six months using the recall method for which also a part of the RUD instrument will be utilized. Next, the amount of time spent in caregiving will be monetized using the opportunity cost method which estimates the value of lost informal caregiver benefits due to spending time on providing informal care. For informal caregivers not active on the labor market wage rates of similar people will be imputed. Basically, productivity loss should be included but given the average high age of informal caregivers it can be expected that productivity loss will have a negligible impact on costs because most of them are retired. Nevertheless, based on the results of mean age and employment status of the included caregivers the researchers will decide to whether or not include productivity loss as a cost. The costs of the intervention will be obtained from the current unit cost per day of Baluchonnage and multiplied by the amount of days the in-home respite care was delivered. Currently the daily cost of Baluchonnage is set at 350€/day covered by charity and 65€/day direct cost for the patient. Additional costs above the fixed daily tariff for Baluchonnage will also be included such as: travel expenses during the respite period and having a pet (5€ extra per day). Additionally, willingness to pay for one day of in-home respite care by Baluchon will be obtained from both study groups using the contingent valuation method (CVM). This method can be defined as a stated preference method for eliciting a monetary value to a health care program. In this trial a closed response format will be used. Finally, for use in the decision analytic model, costs of nursing home placement will be derived from the average daily cost for staying in a nursing home in Belgium at the time of completing secondary endpoint.

Descriptive statistics will be represented to draw a clear profile of the characteristics of study participants. Therefore the mean, percentages and the standard deviations of all continuous variables will be displayed. To determine possible baseline differences between the groups, mean values of baseline characteristics will be compared using independent sample t-tests for continuous variables if normally distributed or by performing Pearson's chi-square test for categorical variables. To help control for bias and confounding statistical techniques such as propensity score matching will be used. Propensity score matching can be seen as a tool to simulate a RCT setting. In this way the observed effect can be considered an unbiased estimate of the real effect. To investigate possible effects of the intervention on the primary and secondary outcomes, analysis of variance will be conducted if the outcome variables are normally distributed. A P-value of 0.05 will be considered as significant. All analyses will be based on intention to treat also taking drop-outs into account and avoiding overestimation of respite care effects. When the intervention is effective a cost-effectiveness analysis in a separate economic evaluation plan will be performed. Also ICERs (Incremental Cost-Effectiveness Ratio) will be calculated for the mean and upper and lower confidence levels of the costs and consequences. To explore uncertainty one-way-sensitivity analysis will be conducted around the ICER and illustrated in a Tornado diagram. Additionally, on all input variables a probabilistic sensitivity analysis, also called Monte Carlo analysis, will be conducted to test robustness of the model. These results will also be illustrated. Finally, the results and the willingness to pay threshold of the Belgian Health Care System will be presented in a cost-effectiveness acceptability curve. To compare time to nursing home placement of persons who use respite care to those who don't, the researchers will use Kaplan-Meier survival curves to illustrate association between the comparison groups. By additionally conducting a log-rank test statistical difference between the groups in time to placement can be found.

ELIGIBILITY:
Inclusion Criteria:

* The study participants are caregiver/care-recipient dyads.
* The caregivers must be informal, meaning that they must not be professional healthcare workers in this caregiving role.
* The caregivers have to identify themselves as the main person responsible for the informal care (primary caregiver).
* Also, the caregivers must speak Dutch or French with some fluency and be able to read and write.
* The care-recipient needs to be diagnosed with dementia based on the criteria of DSM fourth edition (Diagnostic and Statistical Manual of Mental Disorders) and must live in the community.
* Dyads in the control group must never had respite care of the Baluchon type in the past, but be eligible and willing to have it. (On the other hand, dyads from the intervention group who have already received in-home respite from the Baluchon type in the past are still allowed for inclusion.)

Exclusion Criteria:

* Caregivers will be excluded if they have cognitive impairments or severe psychiatric comorbidities.
* Control group dyads who already utilized in-home respite care of the Baluchon type will be excluded.
* Another reason for exclusion in the control group is not willing to consider in-home respite via Baluchon.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 355 (Actual)
Dates: Start 2016-01; Primary Completion 2018-06 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Change in burden of caregivers measured using the Zarit Burden Interview-short version | Assessments over 12 months: T0 = baseline (inclusion), T1 = 14 days after intervention (only intervention group), T3 = T0 + 6 months and T4 = T0 + 12 months.
  Burden will be measured using the Zarit Burden Interview-short version (ZBI) which is a 22-item validated self-report questionnaire developed to examine subjective burden of caregivers of people with dementia.

SECONDARY OUTCOMES:
Health related quality of life measured using the EQ-5D-5L | T0 = baseline (inclusion) and T2 = T0 + 6 months.
  Health related quality of life will be measured using the EQ-5D-5L. The EQ-5D-5L is a valid extension of the 3-level questionnaire. It can be defined as a standardized non-disease specific value-based instrument to describe and value health related quality of life.
Frequency of problematic behaviors in care-recipient (RMBPC) | T0 = baseline (inclusion), T1 = 14 days after intervention (only intervention group), T2 = T0 + 6 months
  To measure the frequency of problematic behaviors in the care-recipient and the reaction of caregivers to these behavioral problems, the Revised Memory and Behavior Problems Checklist (RMBPC) will be used. This validated caregiver self-report measure contains 24 items including three domains (depression, memory-related problems and disruption) and two scales to be answered. One scale measures the frequency of problems behaviors of the recipient and the other measures the reactions of the caregiver to this behavior.
Reaction of caregiver to behavioral problems (RMBPC) | T0 = baseline (inclusion), T1 = 14 days after intervention (only intervention group), T2 = T0 + 6 months
  To measure the reaction of caregivers to behavioral problems of the care-recipient the Revised Memory and Behavior Problems Checklist (RMBPC) will be used.
Intention to institutionalize assessed using Desire To Institutionalize scale | T0 = baseline (inclusion), T1 = 14 days after intervention (only intervention group), T3 = T0 + 6 months and T4 = T0 + 12 months.
  The intention to institutionalize the care-recipient will be assessed using Desire To Institutionalize scale (DTI). This questionnaire contains six yes or no questions each measuring the caregiver's desire to institutionalize the recipient into a nursing home, boarding home or assisted living.
Time to nursing home placement | T3 = T0 + 12 months
  Time to nursing home placement will be obtained by measuring the interval from the date of study enrollment to the date of permanent nursing home placement.
Resource use of the care-recipient measured using the Utilization in Dementia instrument | T0 = baseline (inclusion) and T2 = T0 + 6 months.
  Resource use of the care-recipient will be measured using the Utilization in Dementia instrument (RUD). This valid, standardized and widely used instrument can be used for collecting data on resource use of dementia.

CONTACTS AND LOCATIONS:
Overall Officials: Lieven Annemans, PhD, Study Director — University Ghent
Locations (1):
- Ghent University-Public Health Department, Ghent, East-Flanders, Belgium

REFERENCES:
- [Derived] Vandepitte S, Van Wilder L, Putman K, Van Den Noortgate N, Verhaeghe S, Trybou J, Annemans L. Factors associated with costs of care in community-dwelling persons with dementia from a third party payer and societal perspective: a cross-sectional study. BMC Geriatr. 2020 Jan 16;20(1):18. doi: 10.1186/s12877-020-1414-6. PMID 31948386
- [Derived] Vandepitte S, Putman K, Van Den Noortgate N, Verhaeghe S, Annemans L. Effectiveness of an in-home respite care program to support informal dementia caregivers: A comparative study. Int J Geriatr Psychiatry. 2019 Oct;34(10):1534-1544. doi: 10.1002/gps.5164. Epub 2019 Jul 11. PMID 31243801
- [Derived] Vandepitte S, Van Den Noortgate N, Putman K, Verhaeghe S, Annemans L. Effectiveness and cost-effectiveness of an in-home respite care program in supporting informal caregivers of people with dementia: design of a comparative study. BMC Geriatr. 2016 Dec 2;16(1):207. doi: 10.1186/s12877-016-0373-4. PMID 27912740